CLINICAL TRIAL: NCT02164708
Title: Healthy Student Initiative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: Federal Economic Development Agency for Southern Ontario (Unknown)
Responsible Party: Principal Investigator, Paul Ritvo, Associate Professor, York University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2012 - 170
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Depressive Self-Criticism
Keywords: mindfulness meditation, mental health, self-criticism
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mindfulness Meditation (Experimental): The program progressively trained students in "mindfulness of breathing", a form of meditation frequently employed secularly. The tutorials were held on campus five times weekly, led by a faculty member and a graduate student who were trained, experienced MM practitioners. The tutorials were one hour in duration and typically involved 40-45 minutes of guided MM followed by a question-answer period that addressed recent research findings. Program participation required attendance at one tutorial per week, and participants were encouraged to maintain autonomous MM practice.
  Interventions: Behavioral: Mindfulness Meditation

INTERVENTIONS:
Behavioral: Mindfulness Meditation — The program progressively trained students in "mindfulness of breathing", a form of meditation frequently employed secularly. The tutorials were held on campus five times weekly, led by a faculty member and a graduate student who were trained, experienced MM practitioners. The tutorials were one hour in duration and typically involved 40-45 minutes of guided MM followed by a question-answer period that addressed recent research findings. Program participation required attendance at one tutorial per week, and participants were encouraged to maintain autonomous MM practice.

SUMMARY:
This paper extends prior research by exploring how students with self-critical (SC) traits respond to mindfulness meditation (MM) with a twofold purpose: i) to study anxiety sensitivity and mood changes during the school year as students attended MM tutorials ii) to study the relationship between self-criticism and MM-related benefits over time. This paper reports on participants' mood and anxiety sensitivity changes before, during, and after the MM program and the association between depressed mood and SC levels. Participants were trained in MM over two continuous semesters, with two specific hypotheses guiding evaluations:

1. Participants overall would report progressive improvements in psychological well-being as measured by mood and anxiety sensitivity variables, reflecting the effectiveness of the MM program.
2. Elevations in self-critical personality traits would predict greater improvements in depressed mood, given the greater need to neutralize cognitive events related to negative moods.

DETAILED DESCRIPTION:
A total of 71 undergraduate students in a large public university participated in weekly MM sessions through the Fall & Winter semesters of the 2012/2013 academic year. Recruitment was facilitated through in-class announcements and poster and print advertisements. Online and paper surveys elicited self-report data (reflecting mental health profiles) at program initiation which served as baseline measures for the September-October study period, written informed consent was also obtained during this time. Inclusion criteria included: 1) currently enrolled (part-time-full-time); 2) computer access at the university or elsewhere and/or smartphone access Following a standard within-subjects design, participants were required to complete the psychological measures at 3 additional assessment periods; Time 2 (November-December), Time 3 (January-February), and Time 4 (March-April). To alleviate demands on the students partaking in weekly MM sessions, follow-up assessments were provided in paper and electronic form and completed autonomously. Study participants were given $50 cash payments for full study participation and the study met the ethical guidelines and received approval from the Human Participants Review Subcommittee of the university site where the study was conducted.

The program progressively trained students in "mindfulness of breathing", a form of meditation frequently employed secularly. The tutorials were held on campus five times weekly, led by a faculty member and a graduate student who were trained, experienced MM practitioners. The tutorials were one hour in duration and typically involved 40-45 minutes of guided MM followed by a question-answer period that addressed recent research findings. Program participation required attendance at one tutorial per week, and participants were encouraged to maintain autonomous MM practice.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled (part-time-full-time) OR current staff members at university
* Computer access at the university or elsewhere and/or smartphone access

Exclusion Criteria:

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Profile of Mood States | 6 months
  Inventory to assess mood states

SECONDARY OUTCOMES:
Anxiety Sensitivity | 6 months
  Inventory to assess anxiety sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ritvo, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

REFERENCES:
- [Result] Ritvo, P., Vora, K., Irvine, J., Mongrain, M., Azargive, S., Muhammad Abid, A., … Cribbie, R. (2013). Reductions in Negative Automatic Thoughts in Students Attending Mindfulness Tutorials Predicts Increased Life Satisfaction. International Journal of Educational Psychology, 2(3), 272-296. doi:10.4471/ijep.2013.28